CLINICAL TRIAL: NCT06683248
Title: The Effects of Night Shift Work on Health Across the Menstrual Cycle: a Pilot Study
Brief Title: The Effects of Night Shift Work on Health Across the Menstrual Cycle
Acronym: MENSLEEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Christian Benedict, Senior lecturer, Uppsala University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-04191
Record Dates: First submitted 2024-10-15; First posted 2024-11-12 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Sleep Deprivation; Menstrual Cycle; Brain Health; Metabolism; Microbiota; Immune System
Keywords: Estrogen
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sleep deprivation (Experimental): All participants will undergo an 8-hour sleep opportunity, immediately followed by a night of total sleep deprivation.
  Interventions: Other: Investigate sleep deprivation

INTERVENTIONS:
Other: Investigate sleep deprivation — Sleep deprivation
  Devices used:
  Dreem band for EEG Actiheart Tobii Eye tracker Blood glucose monitor Blood pressure cuff Mira fertility tracker Galvanic skin response K5: wearable metabolic system Fitbit: wearable technology Withings sleep analyzer Body composition monitor

SUMMARY:
The study aims to investigate the effects of sleep deprivation on women's health across different phases of the menstrual cycle.

DETAILED DESCRIPTION:
Modern society demands around-the-clock services, with an estimated 20% of workers involved in night shifts. Shift work disrupts the circadian rhythm and has been linked to increased risks of obesity, metabolic syndrome, glucose dysregulation, and immune system issues. Sleep deprivation, especially during wakeful nights, is associated with elevated levels of central nervous system biomarkers like Tau and Amyloid-β proteins, which are implicated in brain disorders such as Alzheimer's disease.

However, the effects of sleep deprivation on women, particularly in relation to hormonal fluctuations during the menstrual cycle, remain largely unexplored. The menstrual cycle, which occurs in cis-women of childbearing age, involves significant fluctuations in estrogen, a hormone known for its neuroprotective properties. Estrogen impacts memory, executive function, and may play a role in protecting against neurodegenerative conditions like Alzheimer's disease. Previous studies have largely focused on men or women using hormonal contraceptives, leaving a gap in understanding how natural hormonal cycles impact the response to sleep deprivation.

This study addresses this gap by focusing on healthy young women with regular menstrual cycles who do not use hormonal contraceptives. Participants will undergo an adaptation night followed by a sleep condition and a wake condition experiment. The goal is to better understand how hormonal changes throughout the menstrual cycle influence the body's response to sleep deprivation and stress, particularly in areas such as metabolism, brain function, and immune, system, and microbiota.

ELIGIBILITY:
Inclusion Criteria:

- Healthy

Exclusion Criteria:

* Use of hormonal contraceptives
* Chronic disease
* Regular use of nicotine
* Use of medication
* Consumes excessive amounts of alcohol or coffee

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The effect of sleep deprivation vs sleep on brain health across the menstrual cycle | 1 year
  Blood analysis for neurodegenerative biomarkers, specifically Tau protein phosphorylated at amino acid 181 and 231, Aβ40 and Aβ42, GFAP, NfL.
The effects of sleep deprivation across the menstrual cycle on EEG | 1 year
  The Dreem headband will be used to record EEG, assessing wakefulness levels during the sleep deprivation night through spectral power analysis. It will also be used to generate a hypnogram for sleep stage classification.
The effects of sleep deprivation on metabolic function (TEE) | 2 years
  Energy Expenditure is measured with the K5 wearable system to monitor VO₂ and VCO₂ in real-time, assessing total energy expenditure (TEE).
The effects of sleep deprivation on glucose metabolism | 1 year
  Assessed with an Oral Glucose Tolerance Test (OGTT) and continuous blood glucose monitoring.
The effects of sleep deprivation on leptin/adiponectin ratio | 2 years
  Blood analysis to assess the ratio of leptin/adiponectin for metabolic health throughout the menstrual cycle.
The effects of sleep deprivation on vaginal microbiota identification across the menstrual cycle | 2 years
  Identification and comparison of bacterial species composition and diversity (alpha- and beta-diversity)
The effects of sleep deprivation on vaginal microbiota classification across the menstrual cycle | 2 years
  Classification of community state types (CST)
The effects of sleep deprivation on vaginal microbiota across the menstrual cycle | 2 years
  Changes in total phage content
The effect of sleep deprivation on stress response across the menstrual cycle | 2 years
  An auditory paradigm for stress induction will employ eye tracking to monitor changes in pupil dilation.
The effect of sleep deprivation on stress response across the menstrual cycle | 2 years
  Galvanic skin response measures the electrical characteristics or conductance of the skin as an indirect measure of sympathetic autonomic activity using the change of electrical properties of skin measured continuously throughout an auditory paradigm designed to induce stress.
The effect of sleep deprivation on stress response across the menstrual cycle | 2 years
  Heart rate is tracked to assess autonomic responses to stress throughout the auditory paradigm for stress induction.
The effects of sleep deprivation on immune system profiling across menstrual cycle | 3 years
  Human blood samples are analyzed to determine the levels of proangiogenic neutrophils characterized as CD45+CD3-CD19-CD16+CD49d+VEGFR1+. Additionally, the presence of cytotoxic natural killer (NK) cells defined as CD56dim, CD16+, CX3CR1+, CCR7-, CXCR4dim, and CD57+, alongside non-cytotoxic NK cells, which are identified as CD56bright, CD16-, CX3CR1-, CCR7+, CXCR4 high, and CD57-. The cellular populations are expressed as a percentage of CD45+ positive cells, reflecting the total leukocyte population in the blood. To quantify these cell types, the leukocytes are isolated through gradient centrifugation and analyzed using spectral flow cytometry following incubation with two multicolor antibody panels.
  The technique used is FACS, fluorescence-activated cell sorting.
The levels of 6-sulfatoxymelatonin across the menstrual cycle during sleep and sleep deprivation conditions | 2 years
  Urine levels measured 6-sulfatoxymelatonin during both sleep and sleep deprivation condition
The effects of sleep vs sleep deprivation on ABI across the menstrual cycle | 1 year
  Ankle-Brachial Index (ABI) assessed by comparing blood pressure in legs and arms.
The effects of sleep deprivation on palatability across the menstrual cycle | 2 years
  Subjective rating of palatability for food items on a Visual Analogue Scale (VAS).
  Scale Range: 0 to 100, with 0 indicating "not at all palatable" and 100 indicating "extremely palatable." Higher scores indicate greater palatability, potentially signaling increased appeal for certain foods/calories following sleep deprivation, typically viewed as an adverse outcome.
The effects of sleep deprivation on appetite across the menstrual cycle | 2 years
  Blood analysis for leptin/ghrelin ratio
The effects of sleep deprivation on food arousal across the menstrual cycle | 2 years
  Food arousal response will be assessed using an eye tracker to analyze changes in pupil dilation.
The effects of sleep deprivation on hunger across the menstrual cycle | 2 years
  A portion size task is administered to the participant on the morning following both sleep and sleep deprivation conditions to assess hunger. Hunger will be measured by the total caloric content of food portions selected by the participant during the task.
The effects of sleep deprivation on psychomotor vigilance across the menstrual cycle | 2 years
  The Psychomotor Vigilance Task (PVT) is a visual reaction time test used to objectively assess sustained attention and alertness. Participants respond as quickly as possible to visual stimuli, with mean reaction time and the number of lapses (missed responses) serving as key outcome measures that reflect cognitive performance, particularly in conditions like sleep deprivation or fatigue.
The effect of salivary cortisol on sleep vs sleep deprivation across the menstrual cycle | 2 years
  Salivary cortisol samples will be collected during the sleep deprivation night and on the following morning after both sleep and sleep deprivation conditions to investigate cortisol levels in response to sleep loss across menstrual cycle.
Oral microbiota changes across menstrual cycle and sleep deprivation | 4 years
  Analyze the changes in the oral microbiota across the menstrual cycle in sleep and sleep deprivation conditions by investigating shifts in microbial composition, diversity, and the abundance of bacteria. This could provide insights into how sleep patterns and menstrual phases interact to impact oral health.

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided